CLINICAL TRIAL: NCT01365494
Title: A Phase IV, Multi-center, Randomized, Open-label Study of PCECV (Rabipur®) Comparing the Immunogenicity and Safety of Two Different Simulated Post Exposure Schedules (Zagreb 2-1-1 Versus Essen Regimen 1-1-1-1-1) in Healthy Indian Subjects
Brief Title: Immunogenicity and Safety of Rabies Vaccine, Administered With Two Different Simulated Post Exposure Schedules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V49_25
Record Dates: First submitted 2011-05-30; First posted 2011-06-03 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Rabies
Keywords: Rabies; rabies vaccines; post-exposure prophylaxis
MeSH Terms: conditions — Rabies

ARMS (2):
- Group A-Zagreb (Active Comparator): Purified Chick Embryo Cell Inactivated Rabies Vaccine, administered intramuscularly (IM) according to the 2-1-1 (Zagreb) schedule (i.e., 2 doses of vaccine administered on day 0 and 1 dose of vaccine each administered on day 7 and day 21)
  Interventions: Biological: Purified Chick Embryo Cell Inactivated Rabies Vaccine
- Group B-Essen (Active Comparator): Purified Chick Embryo Cell Inactivated Rabies Vaccine, administered IM according to the 1-1-1-1-1 (Essen) schedule (i.e., 1 dose of vaccine administered on day 0, 3, 7, 14, and 28)
  Interventions: Biological: Purified Chick Embryo Cell Inactivated Rabies Vaccine

INTERVENTIONS:
Biological: Purified Chick Embryo Cell Inactivated Rabies Vaccine — Two group (Zagreb and Essen) will receive Rabipur vaccine IM according to either Zagreb or Essen schedules.

SUMMARY:
This study was planned to establish the non-inferiority of Rabipur administered as simulated post exposure Zagreb schedule as compared to Essen schedule, in healthy Indian adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of age ≥ 18 years.
2. Individuals who had given written consent.
3. Individuals in good health and available for all the visits scheduled in the study.

Exclusion Criteria:

1. Pregnancy or unwillingness to practice acceptable contraception.
2. A history of Rabies vaccination.
3. History of allergy to egg protein.
4. Known hypersensitivity to neomycin, tetracycline, amphotericin-B or any other vaccine component.
5. A significant acute or chronic infectious disease or use of antibiotics that may impact the subject's safety and /or immunogenicity in the Investigators opinion at the time of enrolment.
6. Body temperature ≥38.0°C (≥ 100.4°F) within 3 days of study vaccination.
7. Treatment with an anti-malarial drug, up to two months prior to the study.
8. Individuals who received any other vaccines within 28 days prior to enrollment.
9. Subjects who have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks.
10. Any planned surgery during the study period.
11. Subjects who have cancer disorders excluding nonmelanotic skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (3):
- India (3):
  - Kempegowda Institute of Medical Sciences Hospital (KIMS), Bangalore, Karnataka
  - Mandya Institute of Medical Sciences, Mandya, Karnataka
  - Padmashree Dr. D.Y Patil Hospital, Pune, MS

REFERENCES:
- [Derived] Mahendra BJ, Narayana DA, Agarkhedkar S, Ravish HS, Harish BR, Agarkhedkar S, Madhusudana SN, Belludi A, Ahmed K, Jonnalagedda R, Vakil H, Bhusal C, Arora AK. Comparative study on the immunogenicity and safety of a purified chick embryo cell rabies vaccine (PCECV) administered according to two different simulated post exposure intramuscular regimens (Zagreb versus Essen). Hum Vaccin Immunother. 2015;11(2):428-34. doi: 10.4161/21645515.2014.995059. PMID 25692792

RESULTS

PARTICIPANT FLOW:
Groups:
- Zagreb: Rabipur vaccine, administered intramuscularly (IM) according to the 2-1-1 (Zagreb) schedule (i.e., 2 doses of vaccine administered on day 0 and 1 dose of vaccine each administered on day 7 and day 21)
  Purified Chick Embryo Cell Inactivated Rabies Vaccine: Zagreb group received Rabipur vaccine intramuscularly according to either Zagreb schedule.
- Essen: Rabipur vaccine, administered IM according to the 1-1-1-1-1 (Essen) schedule (i.e., 1 dose of vaccine administered on day 0, 3, 7, 14 and 28)
  Purified Chick Embryo Cell Inactivated Rabies Vaccine: Essen group received Rabipur vaccine intramuscularly according to Essen schedule.
Period: Overall Study
Arm/Group | Zagreb | Essen
Started | 126 | 124
Completed | 124 | 121
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Zagreb: Rabipur vaccine, administered intramuscularly (IM) according to the 2-1-1 (Zagreb) schedule (i.e., 2 doses of vaccine administered on day 0 and 1 dose of vaccine each administered on day 7 and day 21)
  Purified Chick Embryo Cell Inactivated Rabies Vaccine: Zagreb group received Rabipur vaccine intramuscularly according to Zagreb schedules.
- Essen: Rabipur vaccine, administered IM according to the 1-1-1-1-1 (Essen) schedule (i.e., 1 dose of vaccine administered on day 0, 3, 7, 14 and 28)
  Purified Chick Embryo Cell Inactivated Rabies Vaccine: Essen group received Rabipur vaccine intramuscularly according to Essen schedules.
- Total: Total of all reporting groups
Arm/Group | Zagreb | Essen | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (8.8) | 27.2 (7.3) | 28.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 58 | 112
  Male | 72 | 66 | 138

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Rabies Virus Neutralizing Antibody (RVNA) Concentration in Each of the Zagreb and Essen Groups on Study Day 14
Description: Immunogenicity was measured as the geometric mean concentrations (GMCs) of rabies virus neutralizing antibody (RVNA) titer , evaluated using the rapid fluorescent focus inhibition test, before vaccination and on study day 14 as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule
Time Frame: On Day 0 and Day 14
Population: Per Protocol Set-All subjects in the FAS (Full analysis set) population who:correctly receive the vaccine, provide evaluable serum sample at day 14, and have no major protocol violation as defined prior to analysis
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- Zagreb: Rabipur vaccine, administered intramuscularly (IM) according to the 2-1-1 (Zagreb) schedule (i.e., 2 doses of vaccine administered on day 0 and 1 dose of vaccine each administered on day 7 and day 21)
  Purified Chick Embryo Cell Inactivated Rabies Vaccine: Zagreb group received Rabipur vaccine intramuscularly according to Zagreb schedule.
Arm/Group | Zagreb | Essen
Number analyzed (Participants) | 124 | 120
IU/mL
  Day 0 | 0.09 [0.076 to 0.11] | 0.099 [0.083 to 0.12]
  Day 14 | 12 [11 to 13] | 12 [11 to 13]
Statistical Analysis 1: Comparison: Zagreb vs Essen; To demonstrate non-inferiority in immune response of the Zagreb postexposure schedule of Rabipur to that of the conventional Essen postexposure schedule at study day 14; Test type: Non-Inferiority or Equivalence — Non-inferiority would be achieved if the lower limit of the two-sided 95% CI of the post vaccination (day 14) ratio of GMCs between the groups (GMCGroup Zagreb / GMCGroup Essen) was greater than 0.667; ANOVA; Ratio of GMCs-Zagreb and Essen at day 14 = 1.03, 95% CI 2-sided [0.89 to 1.19]

2. Secondary Outcome: Percentages of Subjects With Anti-RVNA Titer ≥0.5 IU/mL in Zagreb and Essen Groups at Days 7, 14 and 42
Description: Immunogenicity was measured as the percentage of subjects who achieved anti-RVNA titer ≥0.5 IU/mL, at days 0, 7, 14 and 42 as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedule.
Time Frame: Study day 7, 14 and 42
Population: Full Analysis Set- All subjects in the exposed population who provided at least one evaluable serum sample and as randomized
Measure: Number; unit: Percentages of Subjects
Arm/Group | Zagreb | Essen
Number analyzed (Participants) | 126 | 123
Percentages of Subjects
  Day 0 | 6 [3 to 12] | 9 [5 to 15]
  Day 7(N=125,123) | 74 | 97
  Day 14(N=124,123) | 100 | 100
  Day 42(N=124,121) | 100 | 100

3. Secondary Outcome: Ratio of GMCs in Study Groups (Zagreb/Essen Schedules) on Days 7 and 42 as Measured by RVNA Geometric Mean Concentrations
Description: Immunogenicity was measured as the ratio of GMCs of RVNA titer , evaluated using the rapid fluorescent focus inhibition test, on Days 7 and 42 as per Zagreb (2-1-1) and Essen (1-1-1-1-1) postexposure schedules
Time Frame: Day 0, Day 7, Day 14 and Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU\ml
Groups:
- Zagreb: Rabipur vaccine, administered intramuscularly (IM) according to the 2-1-1 (Zagreb schedule) (i.e., 2 doses of vaccine administered on day 0 and 1 dose of vaccine each administered on day 7 and day 21)
  Purified Chick Embryo Cell Inactivated Rabies Vaccine: Zagreb group received Rabipur vaccine intramuscularly according to Zagreb schedule.
Arm/Group | Zagreb | Essen
Number analyzed (Participants) | 126 | 123
IU\ml
  Day 0 | 0.091 [0.077 to 0.11] | 0.099 [0.084 to 0.12]
  Day 7(N=125,123) | 0.66 [0.55 to 0.78] | 1.74 [1.46 to 2.07]
  Day 14(N=124,123) | 12 [11 to 13] | 12 [11 to 13]
  Day 42(N=124,121) | 15 [14 to 16] | 16 [15 to 17]
Statistical Analysis 1: Comparison: Zagreb vs Essen; Test type: Superiority or Other; ANOVA; Ratio of GMCs-Zagreb and Essen at day 7 = 0.38, 95% CI 2-sided [0.3 to 0.48]
Statistical Analysis 2: Comparison: Zagreb vs Essen; Test type: Superiority or Other; ANOVA; Ratio of GMCs-Zagreb and Essen at day 42 = 0.96, 95% CI [0.86 to 1.07]

4. Secondary Outcome: Percentages of Subjects Reporting Adverse Events (AEs)
Description: Adverse events (AEs) were collected for 7 days following administration of each study vaccination or until time of next vaccination (whichever occurred sooner). All reported SAEs and medically attended AEs or AEs that resulted in the premature withdrawal of subjects during the study were collected throughout the study period and all AEs were unsolicited.
Time Frame: All reported SAEs and medically attended AEs or AEs that resulted in the premature withdrawal of subjects were collected up to 42 days after first vaccination. Adverse events were collected throughout the study period
Population: Safety population- All subjects in the Exposed population who provide post vaccination safety data and as vaccinated (as treated)
Measure: Number; unit: percentages of subjects
Arm/Group | Zagreb | Essen
Number analyzed (Participants) | 126 | 123
percentages of subjects
  Any AEs | 17 | 15
  At least possibly related AEs | 4 | 11
  SAE | 0 | 0
  At least possibly related SAEs | 0 | 0
  Deaths | 0 | 0
  Medically Attended AEs | 0 | 0
  Withdrawal from study due to AE | 0.8 | 0

ADVERSE EVENTS:
Time Frame: All reported SAEs and medically attended AEs or AEs that resulted in the premature withdrawal of subjects were collected up to 42 days after first vaccination.
Arm/Group | Zagreb | Essen
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/123
Other Adverse Events (participants affected / at risk) | 3/126 | 8/123
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zagreb (N=126) | Essen (N=123)
Injection site pain (General disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial